CLINICAL TRIAL: NCT05799209
Title: Reduced Environmental Stimulation Therapy (REST) in Methamphetamine Use Disorder: A Pilot Study
Brief Title: Floatation-REST in Methamphetamine Use Disorder: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-001
Record Dates: First submitted 2023-03-07; First posted 2023-04-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Amphetamine-Type Substance Use Disorder
Keywords: Methamphetamine Use Disorder; Floatation Therapy

STUDY DESIGN:
Intervention Model Description: Participants complete both arms of the study on separate days.
Who Masked: Participant, Care Provider
Masking Description: The investigator and participant are masked to study arm until after the participant completes their baseline assessment visit, at which point they are randomized using a sealed envelope.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Reduced Environmental Stimulation Pool (Experimental): floating supine in a pool for a prescribed amount of time (1 total session lasting 1 hour)
  Interventions: Device: Float Pool
- Zero Gravity Chair (Active Comparator): floating supine in a zero-gravity chair for a prescribed amount of time (1 total session lasting 1 hour)
  Interventions: Device: Float Chair

INTERVENTIONS:
Device: Float Pool — Participant floats supine in a pool of water saturated with Epsom salt in an environment which minimizes stimulation of the nervous system, including reduced light, sound, and pressure on the spinal cord.
  Arms: Reduced Environmental Stimulation Pool
Device: Float Chair — Participant floats supine in a zero-gravity chair in an environment which minimizes stimulation of the nervous system, including reduced light, sound, and pressure on the spinal cord.
  Arms: Zero Gravity Chair

SUMMARY:
This early-stage trial aims to examine the feasibility, tolerability, and safety of Floatation-REST (Reduced Environmental Stimulation Therapy) or an active comparison condition in 50 individuals receiving treatment for Amphetamine-Type Substance Use Disorder.

DETAILED DESCRIPTION:
Methamphetamine Use Disorder (MUD) is associated with a barrage of mental and physical health problems including heightened drug craving/relapse/overdose rates, comorbid mood and anxiety disorders, and cardiovascular dysfunction. Unfortunately, MUD is becoming more prevalent. In the U.S., methamphetamine-related treatment admissions are increasing, as are methamphetamine-related deaths in recent years. Despite this substantial burden, there are currently no FDA approved pharmacological treatments for methamphetamine use disorder.

Recent models of addiction highlight the potential role that negative reinforcement plays in relapse, such that stress and negative affect increase drug craving, thereby increasing the likelihood of future drug seeking behaviors despite negative consequences. Consistent with this model, individuals may persist in methamphetamine use to avoid aversive states such as anxiety, depression, fatigue, and other withdrawal symptoms, a cycle known as negative reinforcement. Floatation-REST (Reduced Environmental Stimulation Therapy is a novel non-pharmacologic intervention that has been shown to reduce anxiety/stress in anxious and depressed individuals. It seems plausible that it may have the potential to lessen these aversive states in methamphetamine users, which may also relate to decreased state drug craving/urges to use. To our knowledge, no studies have tested the feasibility/tolerability and safety of floatation-REST in individuals with methamphetamine-type substance use disorder.

The current study investigates the safety and feasibility/tolerability of a single session of floatation-REST in treatment-seeking individuals with methamphetamine use disorder, relative to an active comparator. In this within-subject crossover design, participants will complete two counterbalanced sessions: one in a floatation pool (Pool-REST), and the other in a floatation chair (Chair-REST). Safety and tolerability will be assessed by self-report questionnaires as well as via pre- and post-session ratings of anxiety, stress, and drug craving. Feasibility will be assessed by intervention adherence rate. Findings from this study will inform the design of future feasibility and efficacy studies as well as mechanistic studies of recovery from methamphetamine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-55 years of age
* Meeting criteria for a primary DSM-5 diagnosis of current methamphetamine use disorder
* Has completed at least two weeks of inpatient treatment (translating into having at least two weeks of drug/alcohol sobriety) at one of the two recruitment sites (Grand Addiction and Recovery Center or Women In Recovery) and is still currently enrolled in this treatment at the time of the study
* Capable of completing all measures during each session of the experiment: able to provide written informed consent and must have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.

Exclusion Criteria:

* Has any of the following DSM-5 disorders: Schizophrenia Spectrum and Other Psychotic Disorders OR Bipolar I Disorder
* Participant fails to adhere to our "Pre-float checklist".
* Any antihistamine that causes drowsiness (e.g., Benadryl).
* Caffeine or nicotine consumed within the past 2 hours.
* Reports a history of unstable liver or renal insufficiency; glaucoma; diabetes; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
* A breathalyzer test positive for alcohol or a drug-positive urine test at either session.
* Non-correctable vision or hearing problems.
* Unwillingness or inability to complete major aspects of the study protocol (e.g., floating). However, failing to complete some individual aspects will be acceptable (e.g., being unwilling to answer individual items on a questionnaire).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Side Effects | Over the span of the intervention, up to two weeks
  As a proxy of safety, the negative and positive side effects reported by each participant is equal to the number of instances during the study when a participant reports elevations above mild for any negative or positive effects on the side effect checklist (administered after each float session)

SECONDARY OUTCOMES:
Completion Rate | Over the ten days of intervention
  As a proxy of feasibility, the rate of adherence for the group is equal to the total randomized minus (dropout plus withdrawn) divided by total randomized
  All participants are given up to 3 opportunities to reschedule missed appointments, after which they are withdrawn from the study.
Stimulant Craving on the Stimulant Craving Questionnaire (STCQ)-Brief | Through completion of the final float session, up to two weeks
  [Average change pre- to post-intervention]
State Anxiety on the State Trait Anxiety Inventory (STAI) | Through completion of the final float session, up to two weeks
  Average change pre to post-intervention
Negative Affect on Positive and Negative Affective Schedule- X | Through completion of the final float session, up to two weeks
  Negative Affect subscale [Average change pre- to post-intervention]
Positive Affect on Positive and Negative Affective Schedule- X | Through completion of the final float session, up to two weeks
  Positive Affect subscale [Average change pre to post-intervention
Fear on Positive and Negative Affective Schedule- X | Through completion of the final float session, up to two weeks
  Fear subscale [Average change pre- to post-intervention]
Fatigue on Positive and Negative Affective Schedule- X | Through completion of the final float session, up to two weeks
  Fatigue subscale [Average change pre- to post-intervention]
Serenity on the Positive and Negative Affect Schedule-X (PANAS-X) | Through completion of the final float session, up to two weeks
  Serenity subscale [Average change pre to post-intervention]
Joviality on the Positive and Negative Affect Schedule-X (PANAS-X) | Through completion of the final float session, up to two weeks
  Joviality subscale [Average change pre to post-intervention]
Attentiveness on the Positive and Negative Affect Schedule-X (PANAS-X) | Through completion of the final float session, up to two weeks
  Attentiveness subscale [Average change pre to post-intervention]

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No